CLINICAL TRIAL: NCT00149916
Title: Multicenter, Open-label Follow-up Study on the Safety of Enteric-coated Mycophenolate Sodium in Renal Transplant Patients.
Brief Title: Follow-up Study of Safety of Enteric-coated Mycophenolate Sodium in Patients Who Successfully Completed Study CERL080A0107
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CERL080A107E
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-11

CONDITIONS: Renal Transplant
Keywords: Renal Transplant, adults, immunosuppressants
MeSH Terms: interventions — Mycophenolic Acid

ARMS (1):
- Mycophenolate sodium (enteric coated) (Experimental)
  Interventions: Drug: Mycophenolate sodium (enteric coated)

INTERVENTIONS:
Drug: Mycophenolate sodium (enteric coated)

SUMMARY:
Aim of study is to provide safety and tolerability data on enteric-coated mycophenolate sodium in regard to adverse events, serious adverse events and patient and graft survival. After successful completion of the study CERL080A0107 study, patients could continue to receive enteric-coated mycophenolate sodium.

ELIGIBILITY:
Inclusion Criteria:

* Cadaveric or living donor kidney transplant recipients who completed the study CERL080A0107

Exclusion Criteria:

* Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2000-04; Primary Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
To assess gastro-intestinal tolerability

SECONDARY OUTCOMES:
Efficacy/safety of enteric-coated mycophenolate sodium based on AE reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis